CLINICAL TRIAL: NCT02486991
Title: Impact of Intramucosal Vertical Incisions on the Coronally Positioned Tunnel Using Acellular Dermal Matrix
Brief Title: Tunnel With and Without Intramucosal Vertical Incisions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Director-Graduate Periodontics Program, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.0532
Record Dates: First submitted 2015-06-19; First posted 2015-07-01 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession | interventions — Alloderm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tunnel + AlloDerm® (Active Comparator): A coronally positioned tunnel (CPT) technique for root coverage will be used alone with acellular dermal matrix (AlloDerm®).
  Interventions: Procedure: Tunnel + AlloDerm®
- Tunnel + AlloDerm® + Verticals (Experimental): The use of intramucosal vertical incisions in addition to a coronally positioned tunnel (CPT) technique for root coverage will be used with acellular dermal matrix (AlloDerm®).
  Interventions: Procedure: Tunnel + AlloDerm®; Procedure: Tunnel + AlloDerm® + Verticals

INTERVENTIONS:
Procedure: Tunnel + AlloDerm® — A coronally positioned tunnel (CPT) technique for root coverage will be used alone with acellular dermal matrix (AlloDerm®).
Procedure: Tunnel + AlloDerm® + Verticals — The use of intramucosal vertical incisions in addition to a coronally positioned tunnel (CPT) technique for root coverage will be used with acellular dermal matrix (AlloDerm®).
  Arms: Tunnel + AlloDerm® + Verticals

SUMMARY:
Thirty patients will be treated: 15 with a coronally positioned tunnel technique plus intramucosal verticals with AlloDerm® (test treatment) and 15 with a coronally positioned tunnel technique alone with AlloDerm® (control treatment). The surgical procedure for the control sites will consist of a coronally positioned tunnel preparation that is a modification of a previous tunnel technique described by Allen AL (Allen AL, 1994a/1994b). This tunnel technique was modified to include coronal positioning of the soft tissue over an allograft (E.P Allen). The surgical procedure for the test sites will consist of a coronally positioned tunnel preparation (E.P. Allen) plus the use of mesial and/or distal intramucosal verticals, a modification of the vestibular incision subperiosteal tunnel access (VISTA) approach (Zadeh H, 2011). Each patient will provide at least one Miller Class I or II facial recession defect, ≥ 3 mm. Patients will be randomly selected by a coin toss to receive either the test or control treatment. Three exams for measurements will be performed per patient on total: preoperative, at week eight and 16 (4 months) postoperatively. The primary aim is to compare the percent root coverage obtained with acellular dermal matrix using the coronally positioned tunnel technique alone or with intramucosal verticals.

DETAILED DESCRIPTION:
Thirty patients will be treated: 15 with a coronally positioned tunnel technique plus intramucosal verticals with AlloDerm® (test treatment) and 15 with a coronally positioned tunnel technique alone with AlloDerm® (control treatment). The surgical procedure for the control sites will consist of a coronally positioned tunnel preparation that is a modification of a previous tunnel technique described by Allen AL (Allen AL, 1994a/1994b). This tunnel technique was modified to include coronal positioning of the soft tissue over an allograft (E.P Allen). The surgical procedure for the test sites will consist of a coronally positioned tunnel preparation (E.P. Allen) plus the use of mesial and/or distal intramucosal verticals, a modification of the vestibular incision subperiosteal tunnel access (VISTA) approach (Zadeh H, 2011). In both the test and control group, the AlloDerm® will be sutured using a continuous sling suture technique with a Maxon 5-0, 3/8 circle 13 mm needle and the tissue will be coronally positioned and sutured separately using a continuous sling suture technique (line angle to line angle) with PTFE 4-0, 3/8 circle 13.1 mm needle. In the test group, the intramucosal vertical incisions will be sutured using simple interrupted sutures with PTFE 4-0, 3/8 circle 13.1 mm needle. Each patient will provide at least one Miller Class I or II facial recession defect, ≥ 3 mm. Each patient will initially receive a full diagnostic work-up to include the periapical and bite-wing radiographs of the selected site and adjacent teeth, study casts, intra-oral photographs, and full mouth clinical examination. Pre-surgical preparation will include detailed oral hygiene instructions, scaling and root planing under local anesthesia, and occlusal adjustment if indicated. Baseline data on test and adjacent teeth will be recorded on the day of surgical treatment to include: Miller's classification of recession defects, Plaque Index, Gingival Index, Bleeding on Probing Index, Gingival Margin Levels (Recession), Keratinized Tissue, Clinical Attachment Level, Clinical Tooth Mobility, Creeping Attachment, Tooth Vitality, Radiographic Examination, Patient Models, and Clinical photos. Patients will be randomly selected by a coin toss to receive either the test or control treatment. Mentor will toss the coin immediately prior to beginning surgical procedure. Patients will be evaluated postoperatively for a period of 4 months. The examiner will be blinded and will not be aware of the patient treatment at any time during the term of the study. Three exams for measurements will be performed per patient on total: preoperative, at week eight and 16 (4 months) postoperatively. The primary aim is to compare the percent root coverage obtained with acellular dermal matrix using the coronally positioned tunnel technique alone or with intramucosal verticals. Means and standard deviations will be calculated for all parameters. Statistical significance of the mean residual recession data for each parameter will be analyzed using a paired t-test to detect within group statistical differences and an unpaired t-test to detect between group statistical differences. The sample size of 15 per group will afford 80% statistical power to detect a difference of 1.0 mm coverage between groups. Sample size and power calculations are based on data from previous studies.

All surgical procedures will be completed by one operator under the direction of one mentor. First, presurgical measurements will be taken. Defect width will be measured horizontally at the interproximal osseous crest level and 1.0 mm coronal to the defect base. Probing depths, width of keratinized tissue, and gingival margin levels will also be measured. Next, treatment modality will be determined and assigned to the defect. Local anesthesia will be administered, tissue elevated, and measurements of the level of the alveolar crest will be made directly in reference to the CEJ. The alveolar crest will be measured vertically from the mid-buccal, or greatest point of the defect, and proximal osseous crest levels. The soft tissue recession defect will be measured horizontally and vertically for the osseous measurements. Root surfaces will be meticulously root planed using hand instruments to obtain a smooth, hard root surface, then the incisions will be made. No osseous recontouring will be performed.

The surgical procedure for the control sites will consist of a coronally positioned tunnel preparation that is a modification of a previous tunnel technique described by Allen AL (Allen AL, 1994a/1994b). This tunnel technique was modified to include coronal positioning of the soft tissue over an allograft (E.P Allen). Split-thickness dissection beyond the mucogingival junction will be made to elevate the tissue and allow adequate coronal positioning. The tunnel is dissected using a specialized microsurgical kit. The tunnel and ADM will extend at least one tooth mesial and distal to the recession site. Papillae are completely elevated off the osseous crest so that the whole tissue complex is mobile and can be coronally positioned. In cases where access is difficult, an incision will be made to release the papilla to prevent tearing the tissue.

The surgical procedure for the test sites will consist of a coronally positioned tunnel preparation (E.P. Allen) plus the use of mesial and/or distal intramucosal verticals, a modification of the vestibular incision subperiosteal tunnel access (VISTA) approach (Zadeh H, 2011). The procedure will begin with one or multiple (mesial and distal) intramucosal vertical incisions, with the location of access depending on the sites being treated. The intramucosal incision is made through the periosteum to elevate a subperiosteal tunnel, exposing the facial osseous plate as well as root dehiscences. The tunnel and ADM will extend at least one tooth mesial and distal to the recession site. The tunnel is dissected using a specialized microsurgical kit. It is crucial to extend the tunnel elevation sufficiently beyond the mucogingival margin as well as through the gingival sulci of the teeth being augmented to allow for low-tension coronal repositioning of the gingiva. The tunnel is extended interproximally under each papilla as far as the embrasure space permits, without making any surface incisions through the papillae.

For both control and test groups, the Alloderm® is hydrated in two baths: first with sterile saline for a minimum of five minutes or until the backing separates from the Alloderm®, the second with sterile saline plus tetracycline at a ratio of 5 mg tetracycline / 1 mL saline until the tissue is fully hydrated. Next, the AlloDerm® will be adjusted to completely cover the defect, positioned against the root surface, at the CEJ, and the inferior and lateral borders of the grafts will extend at least 3.0 mm beyond the osseous defect margins. In the control group, the AlloDerm® will be sutured using a continuous sling suture technique with a Maxon 5-0, 3/8 circle 13 mm needle and the tissue will be coronally positioned and sutured separately using a continuous sling suture technique (line angle to line angle) with PTFE 4-0, 3/8 circle 13.1 mm needle. In the test group, the AlloDerm® will be sutured using a continuous sling suture technique with a Maxon 5-0, 3/8 circle 13 mm needle and the tissue will be coronally positioned and sutured separately using a continuous sling suture technique (line angle to line angle) with PTFE 4-0, 3/8 circle 13.1 mm needle. The intramucosal vertical incisions will be sutured using simple interrupted sutures with PTFE 4-0, 3/8 circle 13.1 mm needle.

Post-operative instructions will be given to the patients along with prescriptions, in appropriate cases, for systemic doxycycline hyclate 100 mg once a day for 14 days; an anti-inflammatory agent (naproxen 375 mg q12h for 7 days); an analgesic (Vicodin ES q6-8h prn pain); a steroid, Medrol dose pack, 21 tablets of 4 mg methylprednisolone; 6 tablets on day 1, 5 on day 2, decrease by 1/day until last tablet dose on day 6, or dexamethazone 1mg, 18 tablets, 3 tablets/day for 1st 3 days, 2/day for the next 3 days, 1/day for the last 3 days (always taken in the morning). The surgical procedures will be documented with clinical photographs.

ELIGIBILITY:
Inclusion Criteria:

* At least one Miller Class I or II mucogingival defect ≥ 3 mm (Miller 1985).
* The mucogingival defect must be on a non-molar tooth.
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Patients with debilitating systemic or diseases that significantly affect the periodontium.
* Patients with a known allergy to any of the materials that will be used in the study, including systemic antibiotics (tetracycline and doxycycline).
* Patients requiring antibiotic prophylaxis.
* Root surface restorations at the site of recession.
* No detectable CEJ
* Patients who fail to maintain oral hygiene levels of at least 80% plaque free surfaces.
* Patients who are pregnant or lactating.
* Patients who use tobacco products (smoking or smokeless tobacco).
* Patients with alcohol abuse problems.
* Patients undergoing long-term steroid therapy.
* History of previous root coverage procedures, graft or GTR, on the test teeth.
* Patients who fail to complete the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percent root coverage | 4 months
  Initial and final recession will be measured from the cementoenamel junction to the gingival margin in millimeters. Root coverage will be determined by the amount of initial recession minus the final recession. Percent root coverage will be determined by root coverage divided by initial recession, multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, MS, Principal Investigator — University of Louisville